CLINICAL TRIAL: NCT04256135
Title: Manual Therapy on Activation of the Descending Pain Inhibitory System in Patients With Knee Osteoarthritis
Acronym: MulliganKnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Associate Profesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0902201803618
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Musculoskeletal Manipulations; Osteoarthritis, Knee
Keywords: Mulligan mobilization; Maitland mobilization; Manual therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: It is an experimental, prospective, parallel and longitudinal double-blind study with elderly patients with knee osteoarthritis
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental mobilization: Mulligan (Experimental): Mobilization will be performed while the patient actively performs knee flexion and/or extension depending on the patient's painful or limited movements. Three series of ten repetitions will be performed.
  Interventions: Other: Mulligan mobilization
- Control mobilization: AP Maitland (Active Comparator): The joint mobilization, will be carried out in the knee with both hands, with displacement of the tibia from the front to the back of the femur in an oscillatory way without pain, will be carried out in blocks of 2 minutes with rests of 30 seconds with a duration of about 6 minutes.
  Interventions: Other: AP Maitland mobilization

INTERVENTIONS:
Other: Mulligan mobilization — Mobilization will be performed while the patient actively performs knee flexion and/or extension depending on the patient's painful or limited movements. Three series of ten repetitions will be performed.
  Arms: Experimental mobilization: Mulligan
Other: AP Maitland mobilization — The joint mobilization, will be carried out in the knee with both hands, with displacement of the tibia from the front to the back of the femur in an oscillatory way without pain, will be carried out in blocks of 2 minutes with rests of 30 seconds with a duration of about 6 minutes.
  Other Names: AP Mobilization
  Arms: Control mobilization: AP Maitland

SUMMARY:
Introduction: Knee osteoarthritis is a clinical syndrome which is characterized by pain. It has been shown to cause changes in the nervous system leading to central sensitization. There are factors involved in this disease such as sex (female) or obesity. The most recommended therapy is physical therapy, but manual therapy is needed to cause changes in central sensitization.

Methods: Experimental, prospective, parallel and longitudinal double-blind study, in which two groups are performed: group A (AP mobilizations) and group B (Mulligan's mobilizations). Different variables and questionnaires were used: pressure pain threshold, temporal summation, pain modulation, central sensitization inventory, WOMAC, Times Up & GO, numerical rating scale, Beck, STAI, kinesiophobia, catastrophism, Barthel and mini- cognitive test

DETAILED DESCRIPTION:
INTRODUCTION Osteoarthritis is a degenerative joint disease characterized by a decrease in joint space due to cartilage loss, subchondral sclerosis and osteophytes. Knee osteoarthritis consist in a clinical syndrome that is identified by the presence of pain and can be associated with radiological and laboratory tests Radiology was incorporated by the American College of Rheumatology as a valuable element in the classification of osteoarthritis. Considering the radiological findings and the presence of pain as sufficient criteria for diagnosis The scale used is that of Kellgren and Lawrence, which has 5 grades ranging from 0 to 4, with the greater the degree, the greater the severity marked by the successive presence of decreased interarticular space, sclerosis, cysts and joint deformities. Despite the radiological findings, 40% of the individuals do not have pain.GA is the most significant cause of pain and limitation in the elderly. The prevalence of this disease in Spain is 46% in women and 21% in men over 45 years. Women and African Americans are at greater risk of suffering from osteoarthritis of the knee. The incidence is higher with increasing age. A very important risk factor in the development and progression of this disease is obesity.

The pain of knee osteoarthritis is a multifactorial phenomenon in which structural, neurophysiological and psychosocial factors are involved. With regard to neurophysiological factors, it has been found that there are inflammatory mediators within the articular cartilage which alter afferent sensory inputs and cause plastic changes in the nervous system leading to central sensitization (CS).

Sensitization is defined as an increased response to a painful stimulus, accentuating the signal in the central nervous system, either by increasing the pain signal or by decreasing the pain inhibition signals.

On the other hand, magnetic resonance studies have shown that patients with gonarthrosis have a higher degree of vigilance and a lower capacity to disconnect pain, related to the abnormal activity of different areas of the brain such as the prefrontal areas, the cingulate cortex, the insula, the amygdala and the nucleus accumbens.

The therapies that have had more evidence are pharmacological, non-pharmacological, surgical, infiltration, physical therapies, and lifestyle changes. Because most have side effects, physical therapy is often advised.

The investigators found studies using multimodal treatments, which aim to look for synergistic effects to achieve a better outcome. But it has been shown that if these treatments do not include manual therapy they do not cause changes in central sensitization.

The hypothesis of the study is that with AP and Mulligan's mobilizations the investigators can activate the downward chain.

Primary Objective To evaluate the effectiveness of joint mobilization versus Mulligan's treatment on the activation of conditioned pain modulation, temporal summation, and generalized and local mechanical hyperalgesia Secondary objective As secondary objectives, we will evaluate the effect of accessory mobilizations versus Mulligan's treatment on disability, functionality, central awareness characteristics and psychosocial aspects.

METHODOLOGY RESEARCH DESIGN It is an experimental, prospective, parallel and longitudinal double-blind study with elderly patients with knee osteoarthritis.

PARTICIPANTS Selection of participants: elderly participants from a resident of the elderly in Comunidad de Madrid, who are informed of the procedure and asked for informed consent.

SAMPLE SIZE The sample size will be calculated by means of the "Gpower 3.0.18." computer program.

RANDOM Randomization will be done through the GraphaPad software (GraphPad Software, Inc CA 92037 USA). Patients who meet the inclusion criteria and have none of the exclusion criteria will be entered into the study and the sample will be randomized to obtain the two groups, in opaque, sealed envelopes: A and B.

MASKING The double-blind criteria are met, in which the subjects participating in the study will not know the group to which they were assigned, as well as the physiotherapist in charge of collecting the variable data.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain diagnosed with osteoarthritis of the knee using the criteria of the American College of Rheumatology
* Low or no response to pain medication for osteoarthritis knee pain.

Exclusion Criteria:

* Suffer from any disorder, syndrome or disease that may cause myofascial or neuropathic pain in the lower limbs, such as lumbar radiculopathy, meralgia paresthetica or saphenous nerve entrapment.
* Infiltration with steroids or local anaesthetics during the year prior to the patient's participation in the study or during follow-up.
* History of previous lower extremity or lumbopelvic surgery.
* Ingestion of substances of abuse that may interfere with treatment.
* Contraindications to perform joint therapy mobilizations.
* Previous diagnosis of myopathy or neuropathy (lumbo-sacral plexus)
* Cognitive deficit manifested in the clinical history (Alzheimer, dementia).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Changes in Mechanical Hyperalgesia | Change from Baseline Mechanical Hyperalgesia at 4th sessions
  To measure the pain thresholds by pressure we use an algometer with a surface area of 1cm2 applying it perpendicularly to the skin with a speed of 1 kg / cm2 / s until the patient indicates that the first sensation of pain appears, ceasing at that moment the pressure made. Three measurements will be recorded with an interval of 30 seconds to avoid a temporal sum effect. The measurement will be taken in a distal region of the ipsilateral carpal long radial extender (a point distal to the carpal long radial extender (5cm distal to the lateral epicondyle)) and in the peripatellar region the standard UDP assessment protocol will be used. In the patellar region two sites will be evaluated (3cm medial and lateral to the midpoint of the lateral and medial patella border). A minimum change of 1.62-1.53 kg / cm2 is required for the result to be clinically significant.
Changes in Temporal Summation | Change from Baseline Mechanical Hyperalgesia at 4th sessions
  First the pressure pain thresholds are measured in the lateral area to the patella. Then 10 consecutive pulses are performed in the same locations to provoke the temporal sum, increasing the pressure by 2kg/s and maintaining it for 1 second (followed by 1 second of rest) in each pulse. The intensity of the pain is evaluated at the 1st, 5th and 10th pulse, by means of a numerical scale of the pain (0 being painless and 10 being the maximum pain imaginable).
Changes in Conditioned pain modulation | Change from Baseline Mechanical Hyperalgesia at 4th sessions
  First, pressure pain stimulus (test stimulus) will be conducted in the lateral area to the patella. Second, occlusion cuff will be inflated around the arm of patient until the patient feeling a painful intensity (conditioned stimulus) of 6/10. Finally, after 30 seconds the stimulus will be done. The difference in the mean value of the initial algometry with the mean value of algometry during the conditioning stimulus will indicate the state of the descending pain inhibitory system.

SECONDARY OUTCOMES:
Central sensitization inventory | Baseline
  It serves to identify the symptoms related to central sensitization. It consists of 25 items that are scored from 0: never to 4: always reaching a maximum score of 100. Results are interpreted as follows: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
  We used the Spanish version which has high reliability and validity.
WOMAC Questionnaire | Baseline
  This questionnaire has 24 items grouped in three scales, being 5 items of pain, 2 items of stiffness and 17 items of functional capacity. The score ranges from 0-96, with the higher the score, the worse the pain and disability indicators are considered. To be clinically significant, a change of 7.9 points is needed in the questionnaire.
Test Time Up & Go | Change from Baseline Mechanical Hyperalgesia at 1 month
  This test assesses the mobility and balance of the elderly person, who sits in a chair with armrests and starts to bidet from the seat, walks 3 meters, and turns around, along the path travelled, until sitting, it starts with a rehearsal, being a valid and reliable test. It is evaluated by means of the seconds, being ≤ 10 Independent mobility, ≤ 20 Mostly independent, 20-29 Variable mobility, ≥ 20 Reduced mobility.
Numerical rating scale (NRS) | Change from Baseline Mechanical Hyperalgesia at 4th sessions
  This scale assesses the intensity of subjective pain in a range of 0-10 in which 0 corresponds to no pain and 10 to the worst pain imaginable. NDE in older people without cognitive impairment has demonstrated acceptable reliability, while the Visual Analogical Scale is not recommended in geriatric patients.
Beck Depression Inventory (BDI) | Baseline
  The level of depressive symptomatology was measured by the Spanish version of the Beck Depression Inventory (BDI-II); a self-report measure that assesses affective, cognitive and somatic symptoms of depression.
Anxiety | Baseline
  The state-trait anxiety inventory (STAI) is a questionnaire that measures trait anxiety (a personality factor that predisposes the patient to suffer from anxiety) and the state of anxiety (environmental factors that protect or generate anxiety). Each of the two sub-scales (trait anxiety and state anxiety) consists of 20 items, ranging from 0 (nothing) to 3 (a lot).
Kinesiophobia | Baseline
  Tampa Scale for Kinesiophobia. To assess the fear of movement and pain-related fear. The 11 items are scored 1-4, with total scores ranging from 11 to 44. The addition of all the points obtained from each of the items results in the level of kinesiophobia, with higher scores indicating greater perceived kinesiophobia
Pain catastrophizing | Baseline
  Pain Catastrophizing Scale (PCS). This tool is a 13-item questionnaire designed to measure the three components of pain-related catastrophizing: rumination, magnification, and helplessness, resulting in a unique score. Each item is responded to on a 5-point scale (0 not at all, 4 all the time) relating the degree to which the individual experiences a thought or feeling of a painful situation.
Barthel | Baseline
  The Barthel Index assesses a person's degree of independence by measuring the performance of ten activities of daily living. With a maximum score of 100 points, with the following interpretation of the data: <20 total dependence, 21-60 severe dependence, 61-90 moderate dependence, 91-99 slight dependence, 100 independence.
Mini-Mental State Examination | Baseline
  It is a neuropsychological assessment to estimate the cognitive impairment that the patient may present. It is divided into 11 sections in which a maximum score of 30 points can be achieved, with the lowest score being the most deteriorated. The cut-off point is 22.

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, Phd, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain